CLINICAL TRIAL: NCT03401684
Title: Assessing the Impact of the Resilient Minds Program in Fire Departments
Brief Title: The Resilient Minds Program in Fire Departments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: McMaster University (Other)
Collaborators: Canadian Mental Health Association, Prince Edward Island (Unknown); Canadian Mental Health Association, British Columbia (Unknown); Canadian Mental Health Association, Vancouver-Fraser (Unknown); Vancouver Fire and Rescue Services (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government); Social Sciences and Humanities Research Council of Canada (Other); University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017-4390-GRA
Record Dates: First submitted 2017-12-20; First posted 2018-01-17 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Trauma; Critical Incident; Mental Illness
Keywords: firefighters; mental resiliency; peer support
MeSH Terms: conditions — Wounds and Injuries; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Resilient Minds (Experimental): Four comprehensive, skill-building learning modules in the areas of psychological trauma, mental health problems, resiliency and workplace stress.
  Interventions: Behavioral: Resilient Minds

INTERVENTIONS:
Behavioral: Resilient Minds — The program is designed: 1) to decrease the risk of developing a stress disorder or other mental illnesses due to workplace incidents and/or unhealthy stress; 2) to mitigate the negative impacts of mental illness and trauma through early recognition and early intervention; 3) to support the public while on the frontline; and 4) to improve the psychological health of fire staff while cultivating resilience and enhancing quality of life.
  Other Names: Mental Resiliency

SUMMARY:
The purpose of the study is to assess the impact of a mental health training program in volunteer and career firefighters.

DETAILED DESCRIPTION:
THE PROBLEM: Firefighters are frequently exposed to distressing events, or critical incidents such as motor vehicle accidents, burnt bodies, failed rescue attempts, threats to one's own life, and completed suicides that can trigger posttraumatic stress reactions. Previous research show that first responders and other public safety personnel report frequent exposure to traumatic events and are at increased risk for mental health illnesses.

THE STUDY OBJECTIVE: To assess the impact of a mental health training program in volunteer and career firefighters.

THE STUDY SAMPLE: 600 firefighters: 300 Prince Edward Island volunteer or career firefighters, 300 Vancouver career firefighters

INTERVENTION: Vancouver Fire & Rescue Services and the Canadian Mental Health Association-Vancouver Fraser co-developed a new program called, "Resilient Minds-Building the Psychological Health of Fire Fighters." The Resilient Minds training will educate firefighters about the effects of trauma, how to recognize signs of mental health illness and how to access support after critical events. It also trains firefighters to recognize mental health and addictions in co-workers and how to facilitate their help-seeking.

OUTCOMES: The impact of the program will be assessed by pre- and post-program surveys, 3-month, 6-month, 12-month follow-up surveys.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* can read, understand, speak English
* career or volunteer firefighters in PEI participating in Resilient Minds program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2018-01-25 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Mental Health Knowledge | 0-12 months
  Survey on mental health knowledge (unit of measure = 5-point Likert Scale, "Agree Strongly" to "Disagree Strongly")
Knowledge Retention | 0-12 months
  Survey on retention of program material (unit of measure = 5-point Likert scale, "Not much" to "A Lot")
Work Stress | 0-12 months
  Survey on factors that contribute to work stress (unit of measure = 5-point Likert scale, "Not at all" to "A Lot")
Impact on support levels | 0-12 months
  Survey on program's impacts on peer supports and organizational culture (unit of measure = 5-point Likert scale, "No, it seems less supportive" to "Yes, it seems quite a bit more supportive")

SECONDARY OUTCOMES:
Self-perceived learning | 0-12 months
  Survey on self-perceived learning about psychological trauma and/or mental health challenges (unit of measure = 4-point Likert scale, "Very true" to "Not true")
Helpfulness of training | 0-12 months
  Survey of helpfulness of training (unit of measure = Yes or No response)
Utilization of training | 0-12 months
  Survey on intent and actual usage of information or skills learned from program (unit of measure = Yes or No response)
Critical incidents exposure and impact | 0 months
  Survey on exposures to difficult or stressful things (unit of measure = ratings of frequency and impact on life)
Resilience | 0-12 months
  Survey on mental resiliency (unit of measure = 5-point Likert scale, "Strongly Agree" to "Strongly Disagree")

OTHER OUTCOMES:
Traumatic Life Events Checklist | 3 months
  Survey on lifetime experience with "difficult or stressful things"
PTSD Checklst | 0-12 months
  Survey on PTSD symptoms over past month
Public Safety Officer Stress | 0-12 months
  Survey on stress from being first responder (past 6 months)
Suicidal Behavioural | 0-12 months
  Survey on suicidal behaviours
Anxiety | 0-12 months
  Survey on anxiety symptoms (past 2 weeks)
Depression | 0-12 months
  Survey on mood symptoms (past 2 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Brazil, MAEd, PhD, Principal Investigator — FIREWELL; R. Nicholas Carleton, PhD, Principal Investigator — University of Regina; Steve Fraser, Principal Investigator — Vancouver Fire & Rescue Services; Joy MacDermid, PhD, Principal Investigator — McMaster University & Western University
Locations (5):
- Canada (5):
  - Vancouver Fire and Rescue Services, Vancouver, British Columbia
  - Charlottetown Fire Department, Charlottetown, Prince Edward Island
  - East River Fire Department, Mount Stewart, Prince Edward Island
  - Crossroads Fire Department, Stratford, Prince Edward Island
  - Summerside Fire Department, Summerside, Prince Edward Island